CLINICAL TRIAL: NCT05301244
Title: The Effect of Laughter Yoga on Nurses Psychological Resilience and Sleep Quality During the Pandemic Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Suheyla YARALI, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: suheylasy
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Laughter Yoga
Keywords: Nurse, laughter yoga
MeSH Terms: interventions — Laughter Therapy; Nurses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Experiment and control groups were not clearly stated in the outcome evaluation. Coded as A-B.The person making the assessment was not informed about this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- laughter yoga practice (Experimental): Laughter yoga practiced by a researcher with a laughter yoga practitioner certificate
  Interventions: Other: laughter yoga for nurses; Other: laughter yoga for nurses-Deep breathing exercises; Other: laughter yoga for nurses-Warm-up exercises; Other: laughter yoga for nurses-Childish games; Other: laughter yoga for nurses-Laughter exercises
- Laughter yoga session parts-1 (Experimental): Deep breathing exercises (5 minutes)
  Interventions: Other: laughter yoga for nurses; Other: laughter yoga for nurses-Deep breathing exercises; Other: laughter yoga for nurses-Warm-up exercises; Other: laughter yoga for nurses-Childish games; Other: laughter yoga for nurses-Laughter exercises
- Laughter yoga session parts-2 (Experimental): Warm-up exercises (10 minutes)
  Interventions: Other: laughter yoga for nurses; Other: laughter yoga for nurses-Deep breathing exercises; Other: laughter yoga for nurses-Warm-up exercises; Other: laughter yoga for nurses-Childish games; Other: laughter yoga for nurses-Laughter exercises
- Laughter yoga session parts-3 (Experimental): Childish games (10 minutes)
  Interventions: Other: laughter yoga for nurses; Other: laughter yoga for nurses-Deep breathing exercises; Other: laughter yoga for nurses-Warm-up exercises; Other: laughter yoga for nurses-Childish games; Other: laughter yoga for nurses-Laughter exercises
- Laughter yoga session parts-4 (Experimental): Laughter exercises (15 minutes)
  Interventions: Other: laughter yoga for nurses; Other: laughter yoga for nurses-Deep breathing exercises; Other: laughter yoga for nurses-Warm-up exercises; Other: laughter yoga for nurses-Childish games; Other: laughter yoga for nurses-Laughter exercises

INTERVENTIONS:
Other: laughter yoga for nurses — The experimental group was divided into three groups as 17-17-16 people. For four weeks, laughter yoga sessions were held between 20.00 and 21.00, 2 days a week for each group. Laughter yoga sessions were held for the 1st group between 20.00-21.00 on Mondays and Thursdays, for the 2nd group between 20.00-21.00 on Tuesdays and Fridays, and for the 3rd group between 20.00-21.00 on Wednesdays and Sundays. The first sessions lasted 45 minutes, every other session 40 minutes.
Other: laughter yoga for nurses-Deep breathing exercises — Deep breathing exercises (5 minutes) Breathing is held for 4-5 seconds after deep inspiration. While the arms are brought to the normal position, exhale slowly and rhythmically. When expressing after deep inspiration, the lips can be pursed as if whistling or exhaled with laughter.
Other: laughter yoga for nurses-Warm-up exercises — Warm-up exercises (10 minutes) Rhythm of 1-2, 1-2-3 is added to increase the energy level even more and synchronize the movements of the group. After a few rhythmic clapping movements, another movement is added. Whisking hands left and right. Then an audible rhythm of ho, ho, ha-ha-ha is added to the clapping gesture. Make eye contact with people in the group and smile at them.
Other: laughter yoga for nurses-Childish games — Childish games (10 minutes) Childlike games are used to help laugh without reason just like a child. The group is motivated by visualizing these games in their minds, raising the arms up in the form of a "Y" letter, and saying "very good (applause), very good (applause), hey" with palms facing the sky.
Other: laughter yoga for nurses-Laughter exercises — Laughter exercises (15 minutes) This section includes a variety of laughter exercises such as greetings, strawberry milk, conductor, bonus, hot soup, lion, aloha, bird, appreciation, laughter lotion, elevator, cream cake, and bursting balloon laughter.

SUMMARY:
This study aimed to determine the effects of laughter yoga on the psychological resilience and sleep quality of active nurses during the pandemic period. Initial stage of labor on randomized controlled birth outcomes and maternal satisfaction. A total of 100 nurses, determined by power analysis, were recruited into the randomized controlled, single-blind clinical study. The study included 2 groups (group A nurses who had active contact with patients diagnosed with or at risk of covid-19, group B: nurses who had active contact with patients diagnosed or at risk of covid-19 and participated in laughter yoga practice. Laughter yoga; immune system It has been proven by experimental studies that there is a connection between antibodies and endorphins, that it has a healing effect, that it accelerates the circulatory system as an adverse effect to stress, and that it has a vasodilation effect in the vessels.

DETAILED DESCRIPTION:
The study data were collected by the researchers using online systems with the snowball method due to the pandemic. The inclusion criteria of the study (not having undergone abdominal surgery in the last three months, not having uncontrolled hypertension, not having glaucoma, hernia, epilepsy, not having received a psychiatric diagnosis-treatment, not having received a diagnosis-treatment for sleep problems, having done laughter yoga before) The study consisted of 100 nurses who agreed to participate in the study. Descriptive features form consisting of 13 questions, Connor-Davidson Resilience Scale (CD-RISC) scale and Pittsburgh Sleep Quality Index (PSQI) were used to collect data. Research data were collected in 3 months. During the study, 4 people from the experimental group (3 people did not attend the sessions regularly, 1 person left voluntarily), 6 people from the control group (he left voluntarily) quit the study. Finally, the research was completed with 90 nurses, 46 of which were in the experimental group and 44 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Not have undergone abdominal surgery in the past three months
* Not have uncontrolled hypertension
* Not have epilepsy
* Not have received a psychiatric diagnosis or treatment
* Working actively during the pandemic period

Exclusion Criteria:

* Not attending sessions regularly

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form (questionnaire) | up to 2 weeks
  The form prepared by the researchers consists of a total of 13 questions, including some demographic characteristics (age, education level, marital status, etc.) and professional characteristics (working years, frequently worked shifts, clinic/unit worked during the epidemic period, etc.) of the nurses.
Connor-Davidson Resilience Scale (CD-RISC)-pre-test | up to 5 weeks
  The scale consists of 25 items and has a 5-point Likert type scoring ranging from 'never true' (0) to 'always true' (4). Scale; It consists of three sub-dimensions, namely perseverance and personal competence, tolerance to negative phenomena, and spiritual inclination, and the total score to be taken from the scale is minimum 0 and maximum 100 points. High scores obtained from the scale indicate high levels of psychological resilience. According to the factor structure, perseverance and personal competence with items 1, 5, 10, 11, 12, 15, 16, 17, 18, 19, 21, 22, 23, 24, 25; Resilience levels can be determined by examining tolerance to negative events with items 4, 6, 7, 8, 13, 14, and moral tendency with items 2, 3, 9, 20. The Cronbach's alpha coefficient of the scale was stated as 0.89. In this study, the Cronbach's alpha coefficient of the scale was calculated as 0.92.
Pittsburgh Sleep Quality Index (PSQI)-pre-test | up to 5 weeks
  In the form consisting of a total of 24 questions, scores of 7 components are obtained. PSQI; It consists of seven sub-components that evaluate subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping pills, and dysfunction during the day. The response of each is scored between 0-3 according to symptom frequency. The sum of the scores of the seven components gives the total PSQI score. The total score obtained varies between 0-21, and high values indicate poor sleep quality and high sleep disturbance level. A total score of 6 or above indicates that the sleep quality is clinically significantly worse. The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.80. In this study, the Cronbach's alpha coefficient of the PSQI Scale was calculated as 0.83.

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC)-post-application testing | up to 5 weeks
  The scale consists of 25 items and has a 5-point Likert type scoring ranging from 'never true' (0) to 'always true' (4). Scale; It consists of three sub-dimensions, namely perseverance and personal competence, tolerance to negative phenomena, and spiritual inclination, and the total score to be taken from the scale is minimum 0 and maximum 100 points. High scores obtained from the scale indicate high levels of psychological resilience. According to the factor structure, perseverance and personal competence with items 1, 5, 10, 11, 12, 15, 16, 17, 18, 19, 21, 22, 23, 24, 25; Resilience levels can be determined by examining tolerance to negative events with items 4, 6, 7, 8, 13, 14, and moral tendency with items 2, 3, 9, 20. The Cronbach's alpha coefficient of the scale was stated as 0.89. In this study, the Cronbach's alpha coefficient of the scale was calculated as 0.92.
Pittsburgh Sleep Quality Index (PSQI)-post-application testing | up to 5 weeks
  n the form consisting of a total of 24 questions, scores of 7 components are obtained. PSQI; It consists of seven sub-components that evaluate subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping pills, and dysfunction during the day. The response of each is scored between 0-3 according to symptom frequency. The sum of the scores of the seven components gives the total PSQI score. The total score obtained varies between 0-21, and high values indicate poor sleep quality and high sleep disturbance level. A total score of 6 or above indicates that the sleep quality is clinically significantly worse. The Cronbach Alpha internal consistency coefficient of the scale was found to be 0.80. In this study, the Cronbach's alpha coefficient of the PSQI Scale was calculated as 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Süheyla Yaralı, Yakutiye, Erzurum, Turkey (Türkiye)